CLINICAL TRIAL: NCT02578407
Title: Pilot Study of Accommodative/Vergence Therapy to Modify Accommodative Function in Children With Myopia
Acronym: ACC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Chen, Head, Operation office of Clinical Research Center Institution of Drug Clinical Trials,Zhongshan Opthalmic Center of Sun Yat-sen University, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015ACC
Record Dates: First submitted 2015-10-10; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Accommodative/Vergence Therapy (Experimental): Accommodative/Vergence Therapy. No drug involved.
  Interventions: Other: accommodative/vergence therapy

INTERVENTIONS:
Other: accommodative/vergence therapy — 12 weekly accommodative/vergence therapies

SUMMARY:
This study aims to determine the treatment effect of accommodative/vergence therapy on myopic children by assessment of accommodative function before and after therapy.

DETAILED DESCRIPTION:
1. Specific aims of the proposed clinical trial:

   1.1 To prove accommodative/vergence therapy (AT) can normalize the accommodative function of myopic children.。 1.2 If the accommodation function of myopic children can be improved with AT therapy, the outcome will supply a basic for a randomized, multi-center clinic trail to determine the effectiveness of AT to slow the progression of myopia.
2. Hypothesis:

Accommodative/vergence therapy can normalize the accommodative functions of 8-12 years old Chinese myopic children.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in the trial must:

1. be within the age range of 8 to 12 years old inclusive;
2. -0.75d to -4.50dspherical equivalent by cycloplegic autorefraction in both eyes
3. astigmatism≤1.5d in both eyes；
4. anisometropia≤1.0d；
5. accommodation lag at near(33cm）in right eye by non-cycloplegic auto- refraction ≧1d;
6. have vision correctable to at least 0.8 or better in each eye.

Exclusion Criteria:

Subjects enrolled in the trial must NOT have:

1. current or prior use of progressive addition lens, bifocals, or contact lenses in either eye( prior or current use of single vision lens allowed)；
2. history of any of the following functional defects: strabismus, amblyopia, nystagmus；
3. history of diabetes or seizures；
4. history of any ocular systemic, or neuro-developmental condition that might influence refractive development；
5. use of ocular or systemic medications known to affect accommodation, such as atropine, pirenzepine, and anti-epileptic medications in recent 3 months；
6. history of any ocular surgery that might influence refractive development；
7. developmental disability, attention deficit hyperactivity disorder(ADHD), or learning disability diagnosis in children that in the investigator's discretion would interfere with office-based treatment；
8. relocation anticipated for 3 years；
9. birth weight lower than 1250 grams（2lbs,12oz）；
10. siblings in the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in lag of accommodation assessed by open-field autorefractor from baseline visit at 6 months after 12 weekly vision therapies | Baseline visit, 7th visit(7 weeks after BL), 13th visit (13 weeks after BL), 14th visit(9months after BL, which is also 6months after vision therapies )
  We will measure the lag of accommodation objectively in right eye at 33 cm by using open-field autorefractor. An average of 10 static measurements will be recorded in spherical equivalent dioptric power.

SECONDARY OUTCOMES:
Change in accommodative amplitude assessed by push-up technique from baseline visit at 6 months after 12 weekly vision therapies | Baseline visit, 7th visit(7 weeks after BL), 13th visit (13 weeks after BL), 14th visit(9months after BL, which is also 6months after vision therapies )
  We will measure the accommodative amplitude in right eye by using push-up technique with the use of Gulden accommodation rule. An average of 3 measurements will be recorded in spherical dioptric power.
Change in accommodative variability assessed by open-field autorefractor from baseline visit at 6 months after 12 weekly vision therapies | Baseline visit, 7th visit(7 weeks after BL), 13th visit (13 weeks after BL), 14th visit(9months after BL, which is also 6months after vision therapies )
  We will measure the level of fluctuation in lag of accommodation at 33 cm objectively by using open-field autorefractor. A 1 minute continuous measurement will be taken in right eye. The unit of measurement is spherical equivalent dioptric power.
Change in accommodative facility assessed by flipper bar method from baseline visit at 6 months after 12 weekly vision therapies | Baseline visit, 7th visit(7 weeks after BL), 13th visit (13 weeks after BL), 14th visit(9months after BL, which is also 6months after vision therapies )
  We will measure the accommodative facility at 40 cm by flipper bar method using a ±2.00 diopters lens flipper. 1 measurement will be taken in right eye. The unit of measurement is cycles per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China